CLINICAL TRIAL: NCT07186127
Title: A Retrospective Evaluation of the Effectiveness of Methotrexate Treatment in Cases of Ectopic Pregnancy With Relative Contraindications
Brief Title: Methotrexate Treatment in Cases of Ectopic Pregnancy With Relative Contraindications
Status: Recruiting | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025/05/01/044
Record Dates: First submitted 2025-08-29; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-07

CONDITIONS: Ectopic Pregnancy
Keywords: Ectopic Pregnancy; Relative Contraindication; Methotrexate; Laparoscopic surgery
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Methotrexate; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1 and group 2: Group 1 with indication for MTX treatment and group 2 with relative indication for MTX treatment
  Interventions: Drug: Drug: Methotrexate (MTX) Patients received methotrexate treatment according to institutional protocols. Dosage and administration routes were recorded retrospectively. For patients who did not respond

INTERVENTIONS:
Drug: Drug: Methotrexate (MTX) Patients received methotrexate treatment according to institutional protocols. Dosage and administration routes were recorded retrospectively. For patients who did not respond — MTX medical treatment Laparoscopic salpingectomy Laparoscopic salpingostomy
  Other Names: surgical treatment

SUMMARY:
Study Description (For Patients, Families, and Healthcare Providers)

Purpose:

The aim of this study is to evaluate the effectiveness and safety of methotrexate treatment in women with ectopic pregnancy who belong to a group for whom this treatment is relatively contraindicated.

Background:

Methotrexate is a medication commonly used in the treatment of ectopic pregnancy (a pregnancy that occurs outside the uterus, usually in the fallopian tube). However, in certain conditions - such as kidney or liver dysfunction - methotrexate use may carry increased risks. These situations are known as relative contraindications. This study will retrospectively examine treatment outcomes in this specific patient population.

Method:

The study will analyze medical records of patients who were previously treated with methotrexate for ectopic pregnancy. No new interventions will be performed. The analysis will be based solely on existing clinical data.

Why Is This Important? The findings of this study may help us better understand the safety limits of methotrexate therapy and guide healthcare providers in managing similar cases in the future.

DETAILED DESCRIPTION:
Background and Justification of the Study Ectopic pregnancy poses a significant risk in terms of maternal morbidity and mortality and accounts for approximately 1-2% of all pregnancies. With the advancement of early diagnostic methods, non-surgical treatment options have become more prominent; among these, systemic methotrexate therapy has emerged as a safe and effective alternative, particularly in selected patients. However, when selecting patients for methotrexate treatment, both absolute and relative contraindications that may affect treatment success must be carefully evaluated.

In the literature, data on the use of methotrexate in patients with relative contraindications are limited, and findings regarding treatment response, the rate of transition to surgery, and complications in this patient group remain unclear. This lack of clarity can lead to uncertainty in clinical decision-making.

In this study, the retrospective data of 238 patients diagnosed with ectopic pregnancy and treated with methotrexate at our institution, a training and research hospital, between 2019 and 2024 will be analyzed. The number of patients with relative contraindications and the criteria by which they were deemed eligible for methotrexate treatment will be determined during the analysis phase.

This retrospective observational study aims to identify the factors affecting treatment success, particularly in the group of patients with relative contraindications, thereby contributing to patient selection and management processes. By providing real-world data on current clinical practice, this research may also serve as a foundation for future prospective studies.

Purpose of the Study The aim of this study is to retrospectively examine the clinical data of patients who were treated with methotrexate for ectopic pregnancy at a training and research hospital between 2019 and 2024, in order to evaluate treatment response rates and the factors affecting treatment success. In particular, by analyzing the effectiveness of methotrexate therapy in patients with relative contraindications, the rate of transition to surgical intervention, and complications arising during treatment, the study aims to more clearly determine the suitability of medical treatment for this patient group.

The hypothesis of the research is that methotrexate treatment may be effective and safe in ectopic pregnancy cases that meet appropriate criteria, even in the presence of relative contraindications. In addition, certain clinical and laboratory parameters-such as initial beta-human chorionic gonadotropin (β-hCG) levels, mass size, and the presence of fluid in the recto uterine pouch (Douglas pouch)-are anticipated to play a significant role in predicting treatment success.

Study Protocol Plan Ethics approval for this study was obtained on May 15, 2025. This study is a retrospective, descriptive, and observational analysis conducted at a training and research hospital, evaluating the data of patients who received methotrexate treatment for ectopic pregnancy between 2019 and 2024. Clinical data of a total of 236 ectopic pregnancy cases treated with methotrexate will be assessed by reviewing the hospital information management system and patient records.

The study will include both patients who responded to methotrexate treatment and those who did not benefit from it and required surgical intervention. Detailed evaluations will be conducted on each patient's demographic characteristics, obstetric history, mode of delivery, history of previous ectopic pregnancy, methotrexate dosage and administration method, revision curettage procedures performed during treatment, laboratory findings such as complete blood count (CBC) and beta-human chorionic gonadotropin (β-hCG), ultrasound findings including the identified ectopic focus and the presence of free fluid in the recto uterine pouch (Douglas pouch), treatment duration, length of hospital stay, need for surgical intervention, time taken for β-hCG levels to become negative, and pre- and postoperative β-hCG levels in surgical cases.

Response to methotrexate treatment will be defined as observing the expected decline in β-hCG levels over time and the completion of the process without the need for surgical intervention. Characteristics of patients who did not respond to treatment and required surgery will be analyzed separately to identify potential predictors of treatment failure. Data will be analyzed using Statistical Package for the Social Sciences (SPSS), and in addition to descriptive statistics, significance tests will be applied to evaluate the relationship between various parameters and treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ectopic pregnancy
* Received methotrexate (MTX) treatment
* Underwent surgical treatment due to lack of response to MTX therapy
* Compliant with treatment follow-up

Exclusion Criteria:

* Participants with contraindications to methotrexate (MTX) treatment
* Participants non-compliant with follow-up

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study includes only pregnant women.
Study Population: Patients diagnosed with ectopic pregnancy and treated with methotrexate
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum β-hCG levels (IU/L) | Days 0, 4, and 7 after methotrexate administration
  Serum beta-human chorionic gonadotropin levels measured via blood test on days 0, 4, and 7 of methotrexate treatment.

SECONDARY OUTCOMES:
Hospital stay duration (days) | The duration from treatment initiation to discharge for each patient.
  Number of days each patient remained hospitalized from treatment initiation to discharge.
endometrial thickness (mm), ectopic focus size (mm), and douglas pouch fluid (mm) | DAY 1
  Measured via transvaginal ultrasound at diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: gülhan özüm, md, Principal Investigator — Sağlık Bilimleri Üniversitesi, Bağcılar Eğitim ve Araştırma Hastanesi
Locations (1):
- University of Health Sciences, Training and Research Hospital, Istanbul, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared upon reasonable request after publication, following institutional and ethical guidelines.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 01.05.2025-01.05.2026
Access Criteria: Individual participant data (IPD) will be shared upon reasonable request after publication, following institutional and ethical guidelines. They can be accessed by contacting the principal investigator.

REFERENCES:
- [Result] Cohen A, Bar-On S, Cohen Y, Sandel O, Fouks Y, Michaan N, Tzur T, Levin I. Ruptured ectopic pregnancies following methotrexate treatment: clinical course and predictors for improving patient counseling. Reprod Sci. 2022 Apr;29(4):1209-1214. doi: 10.1007/s43032-022-00881-7. Epub 2022 Feb 14. PMID 35157263

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT07186127/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT07186127/ICF_001.pdf